CLINICAL TRIAL: NCT06512363
Title: A Randomized, Double-blind, Multicenter, Placebo-controlled, Parallel-group, Phase 3 Clinical Study to Investigate the Efficacy and Safety of Ramelteon in Chinese Patients With Chronic Insomnia
Brief Title: A Study of Ramelteon in Chinese Patients With Chronic Insomnia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LMTAP2022-III
Record Dates: First submitted 2024-07-09; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Chronic Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ramelteon 8 mg QN (Experimental)
  Interventions: Drug: Ramelteon
- Placebo (Placebo Comparator)
  Interventions: Drug: Ramelteon placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 8 mg, tablets, orally, once nightly for up to 5 weeks.
  Arms: Ramelteon 8 mg QN
Drug: Ramelteon placebo — Ramelteon placebo-matching tablets, orally, once nightly for up to 5 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Ramelteon in chinese patients with chronic insomnia.

Efficacy will be evaluated on objective and subjective sleep parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years old.
* Chronic insomnia disorder diagnosed according to International Classification of Sleep Disorders, Third Edition, Text Revision (ICSD-3-TR) criteria.
* Self-reported history of all the following on at least 3 nights per week within 4 weeks prior to screening: subjective sleep latency (sSL) greater than or equal to 30 minutes, and subjective total sleep time (sTST) less than or equal to 6.5 hours per night.
* Meeting all the following sleep parameters on the 2 PSG nights during the run-in period: mean latency to persistent sleep (LPS) ≥ 20 min (with neither of the two nights < 15 min), and mean wake after sleep onset (WASO) ≥ 30 min (with neither of the two nights < 20 min).
* Usual bedtime between 20:30 and 01:00, and regular time in bed between 6.5 and 9 h.
* Insomnia Severity Index score≥15 at screening and on Day 1 of the treatment period.
* Understand the study procedures and methods, voluntarily participate in this trial, and sign the informed consent.

Exclusion Criteria:

* Use of ramelteon within 30 days prior to screening.
* Previous non-responders to melatonin receptor agonist therapy.
* Known hypersensitivity to ramelteon or related compounds, including melatonin.
* Sleep schedule changes required by employment (e.g. shift worker), or has flown across greater than three time zones (mainland China is considered as 1 time zone) within 30 days prior to screening and during the study period; or special professionals who need to operate machinery during the study period, such as professional drivers, high-altitude operators, etc.
* Participated in a weight loss program or has substantially altered their exercise routine within 30 days prior to screening and during the study period.
* Previous history of nervous system disorders such as epilepsy, schizophrenia, bipolar mental disorder, neurodevelopmental retardation, and cognitive disorder, or previous history of other mental illness that may affect the safety of the subjects or interfere with the study assessments in the opinion of the investigator.
* Previous history of other sleep disorders secondary to other diseases including moderate to severe obstructive sleep apne, circadian rhythm sleep disturbances, paroxysmal sleeping sickness, and restless legs syndrome.
* Apnea-hypopnea index (AHI) and periodic limb movement index (PLMI) > 15 times/hour detected by PSG monitoring during the run-in period.
* Have previous complex sleep behaviors, such as sleep driving, sleep eating, and sleep phone calls.
* Hamilton Anxiety Scale (HAMA) score ≥ 14 and Hamilton Depression Scale (HAMD) score ≥ 18 at screening.
* Have serious diseases of cardiovascular system, digestive system, respiratory system, urinary system, endocrine system, immune system, etc., which are not suitable for the study judged by the investigators.
* AST or ALT > 3 × ULN, and TBIL > 2 × ULN.
* Patients with HIV or syphilis infection.
* Use of any hypnotics, antidepressants, antipsychotic drugs, anticholinergics, memory-enhancing drugs, antihistamines, centrally acting analgesics, centrally acting muscle relaxants, central nervous system stimulants, strong CYP1A2 inhibitors, strong CYP2C9 inhibitors, strong CYP3A4 inhibitors, strong CYP inducers, or any other therapies for insomnia disorder within 1 week prior to the run-in period or within 5 half-lives of the investigational product, whichever is longer.
* Requirement of taking any prohibited medication during study period.
* History of drug abuse within 1 year prior to screening, or positive urine drug screening.
* History of alcohol abuse within 1 year prior to screening, or unwilling to follow alcohol restriction during the study period.
* Regular daily consumption of excessive tea and coffee drinks, or unwilling to follow tea/coffee restriction during the study period.
* History of smoking addiction or unwilling to follow tobacco restriction during the study period.
* Participated in any other investigational study and taken any investigational drug within 1 month or 5 half-lives prior to screening, whichever is longer.
* Pregnant or lactating women, or planning to have children or both men of reproductive potential and women of childbearing potential disagree to use ≥1 effective contraception throughout the study and within 3 months after the end of the study.
* MEQ-19 score ≤ 49.
* Other conditions that are not considered appropriate by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean Latency to Persistent Sleep Assessed by Polysomnography | Week 1

SECONDARY OUTCOMES:
Mean Latency to Persistent Sleep Assessed by Polysomnography | Week 5
Total Sleep Time Assessed by Polysomnography | Weeks 1 and 5
Sleep Efficiency Assessed by Polysomnography | Weeks 1 and 5
Awake Time after Persistent Sleep Assessed by Polysomnography | Weeks 1 and 5
Number of Awakenings after Persistent Sleep Assessed by Polysomnography | Weeks 1 and 5
Subjective Sleep Latency Assessed by Sleep Diary Questionnaire | Weeks 1, 3 and 5
Subjective Total Sleep Time Assessed by Sleep Diary Questionnaire | Weeks 1, 3 and 5
Subjective Sleep Quality Assessed by Sleep Diary Questionnaire | Weeks 1, 3 and 5
Subjective Awake Time Assessed by Sleep Diary Questionnaire | Weeks 1, 3 and 5
Subjective Number of Awakenings Assessed by Sleep Diary Questionnaire | Weeks 1, 3 and 5
Subjective Ease of Falling Back to Sleep Assessed by Sleep Diary Questionnaire | Weeks 1, 3 and 5
Insomnia Severity Index Score Assessed by ISI Questionnaire | Weeks 3 and 5